CLINICAL TRIAL: NCT07039695
Title: Evaluation of Union Rate of Scaphoid Non-Union Fracture in Adults by Herbert Screw Versus Volar Buttress Plate
Brief Title: Union Rate of Scaphoid Non-Union Fracture in Adults by Herbert Screw Versus Volar Buttress Plate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Khaled Karam Abed El-Aleem Mohammed, Assistant Lecturer of Orthopedic Surgery, Faculty of Medicine, Helwan University, Egypt., Helwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-2020
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Union; Scaphoid; Non-Union Fracture; Herbert Screw; Volar Buttress Plate
MeSH Terms: conditions — Fractures, Ununited

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volar buttress plate group (Experimental): Patients will be treated by a volar buttress plate.
  Interventions: Procedure: Volar buttress plate
- Herbert screw group (Experimental): Patients will be treated by Herbert screw.
  Interventions: Procedure: Herbert screw

INTERVENTIONS:
Procedure: Volar buttress plate — Patients will be treated by a volar buttress plate.
  Arms: Volar buttress plate group
Procedure: Herbert screw — Patients will be treated by Herbert screw.
  Arms: Herbert screw group

SUMMARY:
This study aimed to evaluate the short-term results of treating non-united scaphoid waist fractures with a humpback deformity by graft and internal fixation using a volar buttress plate versus the use of a Herbert screw.

DETAILED DESCRIPTION:
Scaphoid fracture is the most common fracture, accounting for roughly 60% of the total carpal bone fractures and 11 % of all hand fractures.

Nonunion occurs in approximately 5% to 25 % of scaphoid fractures. The scaphoid nonunion will collapse into a humpback deformity, and the lunate, together with the proximal pole, into a dorsal intercalated segment instability, which might end in an advanced carpal collapse.

A scaphoid screw acts to prevent bending at the fracture site with three-point fixation within the cancellous bone of the scaphoid. The proximal and distal points of purchase are achieved by the capture of the screw threads in the cancellous bone of the proximal and distal poles of the scaphoid. The third point occurs within the cancellous bone of the scaphoid waist.

ELIGIBILITY:
Inclusion Criteria:

* Age of a patient is between 20 years to 50 years.
* Non-union or delayed union scaphoid wrist fracture (more than 3 months).
* Closed fracture.
* Patients without previous scaphoid surgery.
* Patients without abnormal renal and/or liver functions.
* Patients without hypocalcemia and/or vitamin D3 deficiency.

Exclusion Criteria:

* Open fracture.
* Patients with proximal or distal fracture of the scaphoid.
* Patients with avascular necrosis of scaphoid.
* Patients with mid-carpal arthritis or pan-carpal arthritis.
* Patients with carpal instability.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Mayo Wrist Score | 3 months post-procedure
  The Mayo Wrist Score is a fast and simple tool comprising four questions that assess pain intensity, wrist function, range of motion, and grip strength. Mayo Wrist Score ranges from 0 to 100. Scores of 90-100 are considered excellent, 80-90 good, 60-80 satisfactory, and below 60 poor.

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) score | 3 months post-procedure
  The Disabilities of the Arm, Shoulder and Hand (DASH) is a 30-item patient-reported outcome measure utilized to assess symptoms and function of the entire upper extremity. The score is calculated on a scale score ranging from 0 (no disability) to 100 (most severe disability).

CONTACTS AND LOCATIONS:
Locations (1):
- Helwan University, Helwan, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.